CLINICAL TRIAL: NCT01448733
Title: A Pilot Study to Evaluate the Safety and Tolerability of CeraVe® Lotion Followed by Fixed Dose Clindamycin Phosphate 1.2% / Benzoyl Peroxide 2.5% Gel in the Morning in Combination With CeraVe® Lotion Followed by Tretinoin 0.05% Gel in the Evening for the Treatment of Facial Acne Vulgaris.
Brief Title: Safety and Tolerability of Acanya Gel in Combination With Atralin Gel for Acne Vulgaris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zeichner, Joshua, M.D. (Individual)
Responsible Party: Principal Investigator, Joshua Zeichner, Director of Cosmetic and Clinical Research, Mt Sinai Dermatology, Zeichner, Joshua, M.D.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Coria Combo
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide; clindamycin phosphate; Gels; Acanya Gel; Atralin Gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acanya Plus Atralin (Experimental): A single, open-label arm treating acne with Cerave lotion plus Acanya gel in the morning in combination with Cerave lotion plus Atralin gel in the evening.
  Interventions: Drug: Benzoyl peroxide 2.5%/clindamycin phosphate 1.2% in the morning with with tretinoin 0.05% gel in the evening

INTERVENTIONS:
Drug: Benzoyl peroxide 2.5%/clindamycin phosphate 1.2% in the morning with with tretinoin 0.05% gel in the evening — Green pea sized amount of Benzoyl peroxide 2.5%/clindamycin phosphate 1.2% in the morning in combination with a green pea sized amount of tretinoin 0.05% gel in the evening
  Other Names: Acanya Gel; Atralin Gel

SUMMARY:
The purpose of this study is to evaluate whether Cerave lotion followed by Acanya Gel in the morning in combination with Cerave lotion followed by Atralin gel in the evening is safe and effective for the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 12 years old.
* Subjects must be in good general health as confirmed by medical history and physical examination.
* Females of child-bearing potential must have a negative urine pregnancy test at the baseline visit and agree to be abstinent or use adequate birth control during the study (oral contraceptives, Norplant, Depo-Provera, or double barrier methods (e.g., condom and spermicide).
* Clear diagnosis of facial acne vulgaris for at least 6 months.
* Subject must have a static Physician's Global Assessment (PGA) of 2 (mild severity) or 3 (moderate severity).
* Disease must be stable or slowly worsening for more than one week prior to entering the study.
* Subjects or their guardians must be able to read, sign, and date the informed consent, and abide by study restrictions for its duration.

Exclusion Criteria:

* Females who are pregnant, attempting to conceive, or breastfeeding.
* Subjects with known hypersensitivity to any ingredients in the study drugs.
* Subjects with overt signs of skin atrophy, telangiectasias or other skin findings that would affect efficacy evaluation.
* Subjects with a current active skin malignancy or infection.
* Subjects requiring the use of medications known to alter the course of acne vulgaris during the study treatment.
* Subjects who have received systemic antibiotics within 2 weeks.
* Subjects using systemic corticosteroids or immunosuppressants within 28 days of entering the study.
* Subjects who have received any topical therapies for acne vulgaris within 7 days of entering the study.
* Subjects taking birth control pills used solely for acne control.
* Subjects who are currently participating in or, within the previous 28 days, have participated in another study for the treatment of acne vulgaris.
* Subjects with clinical conditions that may post a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.
* Subjects who have Crohn's disease, colitis, or if subjects ever developed colitis or severe diarrhea with past antibiotic use.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Cutaneous Tolerability of Combination Therapy of Acanya Gel with Atralin Gel for the treatment of acne vulgaris | 12 weeks
  Evaluation of skin erythema, scaling, drying, and stinging/burning

SECONDARY OUTCOMES:
Efficacy of Combination Therapy of Acanya Gel with Atralin Gel for the treatment of acne vulgaris | 12 weeks
  Evaluation of efficacy as defined as a global assessment of clear or almost clear after 12 weeks of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Mt Sinai Hospital, Department of Dermatology, New York, New York, United States